CLINICAL TRIAL: NCT04697160
Title: An Observational Retrospective Cohort Study of Systemic Therapies for Relapsed or Refractory Diffuse Large B Cell Lymphoma (R/R DLBCL), to Compare Outcomes to Those From Tafasitamab + Lenalidomide in the L-MIND Study
Brief Title: Observational Retrospective Cohort Study of Systemic Therapies for R/R DLBCL
Acronym: RE-MIND2
Status: Completed | Type: Observational
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Other Study IDs: MOR208C213
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received systemic therapies for R/R DLBCL

SUMMARY:
To compare the efficacy outcomes of the L-MIND cohort with the effectiveness in a matched patient population treated with systemic NCCN/ESMO guideline listed regimens administered in routine clinical care.

DETAILED DESCRIPTION:
This retrospective observational cohort study aims to generate a historical control consisting of R/R DLBCL patients who received currently guideline recommended therapies.

ELIGIBILITY:
Eligibility Criteria:

1. Age ≥ 18 years at the initial DLBCL diagnosis.
2. One of the following histologically confirmed diagnosis: DLBCL not otherwise specified (NOS); T-cell/histiocyte rich large B-cell lymphoma (THRLBCL); Epstein-Barr virus (EBV) positive DLBCL of the elderly (EBV-positive DLBCL), Grade 3b Follicular Lymphoma (FL), Composite lymphoma with a DLBCL component with a subsequent DLBCL relapse, according to the Revised European American Lymphoma/World Health Organization (REAL/WHO) classification. Additionally, patients with the evidence of histological transformation to DLBCL from an earlier diagnosis of low grade lymphoma (i.e., an indolent pathology such as FL, marginal zone lymphoma, chronic lymphocytic leukemia) into DLBCL with a subsequent DLBCL relapse are also eligible.
3. Relapsed or refractory DLBCL and received at least 2 systemic regimens for the treatment of DLBCL, including at least 1 anti-CD20 containing therapy.

Non-Eligibility Criteria:

1. Patients with central nervous system (CNS) involvement by lymphoma at initial DLBCL diagnosis.
2. Patients who were treated with CD19-targeted therapy or immunomodulatory drugs (IMiDs) (e.g., thalidomide, LEN) as a frontline DLBCL therapy.
3. Patients who underwent an allogeneic stem cell transplant.
4. Patients who had a prior history of malignancies other than DLBCL, unless the patient has been free of the disease for ≥5 years prior to inclusion.

   Note: Patients with the following malignancies within the 5 years period are still eligible:
   1. basal cell carcinoma of the skin
   2. squamous cell carcinoma of the skin
   3. carcinoma in situ of the cervix
   4. carcinoma in situ of the breast
   5. carcinoma in situ of the bladder
   6. incidental histological finding of prostate cancer (Tumor/Node/Metastasis [TNM] stage of T1a or T1b)
5. Patients who received tafasitamab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed or refractory DLBCL
Sampling Method: Non-Probability Sample
Enrollment: 3573 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Overall/Objective Response Rate (ORR) | through study completion, an average of 1 year
Complete Response Rate (CR) | through study completion, an average of 1 year
Duration of Response (DoR) | through study completion, an average of 1 year
Event Free Survival (EFS) | through study completion, an average of 1 year
Progression Free Survival (PFS) | through study completion, an average of 1 year
Time to next treatment (TTNT) | through study completion, an average of 1 year
Treatment discontinuation rate due to adverse events | through study completion, an average of 1 year
Duration of treatment exposure | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eva Waltl, Study Director — MorphoSys AG
Locations (149):
- United States (21):
  - MorphoSys Research Site, Scottsdale, Arizona
  - MorphoSys Research Site, Clovis, California
  - MorphoSys Research Site, Los Angeles, California
  - MorphoSys Research Site, Orange, California
  - MorphoSys Research Site, Torrance, California
  - MorphoSys Research Site, Broomfield, Colorado
  - MorphoSys Research Site, Chicago, Illinois
  - MorphoSys Research Site, Skokie, Illinois
  - MorphoSys Research Site, Indianapolis, Indiana
  - MorphoSys Research Site, Wichita, Kansas
  - MorphoSys Research Site, Ann Arbor, Michigan
  - MorphoSys Research Site, Minneapolis, Minnesota
  - MorphoSys Research Site, Rochester, Minnesota
  - MorphoSys Research Site, Jackson, Mississippi
  - MorphoSys Research Site, Morristown, New Jersey
  - MorphoSys Research Site, New York, New York
  - MorphoSys Research Site, Charlotte, North Carolina
  - MorphoSys Research Site, Portland, Oregon
  - MorphoSys Research Site, Nashville, Tennessee
  - MorphoSys Research Site, Salt Lake City, Utah
  - MorphoSys Research Site, Spokane, Washington
- Australia (9):
  - MorphoSys Research Site, Adelaide
  - MorphoSys Research Site, Benowa
  - MorphoSys Research Site, Concord
  - MorphoSys Research Site, Darlinghurst
  - MorphoSys Research Site, East Melbourne
  - MorphoSys Research Site, Fitzroy
  - MorphoSys Research Site, Frankston
  - MorphoSys Research Site, Kingswood
  - MorphoSys Research Site, Nedlands
- Austria (6):
  - MorphoSys Research Site, Leoben
  - MorphoSys Research Site, Linz
  - MorphoSys Research Site, Salzburg
  - MorphoSys Research Site, Sankt Pölten
  - MorphoSys Research Site, Vienna
  - MorphoSys Research Site, Wels
- Canada (2):
  - MorphoSys Research Site, Edmonton
  - MorphoSys Research Site, Montreal
- MorphoSys Research Site, Aalborg, Denmark
- France (29):
  - MorphoSys Research Site, Albi
  - MorphoSys Research Site, Amiens
  - MorphoSys Research Site, Angers
  - MorphoSys Research Site, Caen
  - MorphoSys Research Site, Carcassonne
  - MorphoSys Research Site, Castres
  - MorphoSys Research Site, Chambéry
  - MorphoSys Research Site, Grenoble
  - MorphoSys Research Site, La Roche-sur-Yon
  - MorphoSys Research Site, Lille
  - MorphoSys Research Site, Montpellier
  - MorphoSys Research Site, Narbonne
  - MorphoSys Research Site, Nice
  - MorphoSys Research Site, Nîmes
  - MorphoSys Research Site, Orléans
  - MorphoSys Research Site, Paris
  - MorphoSys Research Site, Perpignan
  - MorphoSys Research Site, Pessac
  - MorphoSys Research Site, Pierre-Bénite
  - MorphoSys Research Site, Quimper
  - MorphoSys Research Site, Rodez
  - MorphoSys Research Site, Rouen
  - MorphoSys Research Site, Saint-Brieuc
  - MorphoSys Research Site, Saint-Priest-en-Jarez
  - MorphoSys Research Site, Saint-Quentin
  - MorphoSys Research Site, Toulouse
  - MorphoSys Research Site, Tours
  - MorphoSys Research Site, Troyes
  - MorphoSys Research Site, Vandœuvre-lès-Nancy
- Germany (31):
  - MorphoSys Research Site, Aschaffenburg
  - MorphoSys Research Site, Augsburg
  - MorphoSys Research Site, Bad Liebenwerda
  - MorphoSys Research Site, Cologne
  - MorphoSys Research Site, Donauwörth
  - MorphoSys Research Site, Dresden
  - MorphoSys Research Site, Flensburg
  - MorphoSys Research Site, Frechen
  - MorphoSys Research Site, Freiburg im Breisgau
  - MorphoSys Research Site, Göttingen
  - MorphoSys Research Site, Halle
  - MorphoSys Research Site, Hamburg
  - MorphoSys Research Site, Hanover
  - MorphoSys Research Site, Heidelberg
  - MorphoSys Research Site, Heilbronn
  - MorphoSys Research Site, Landshut
  - MorphoSys Research Site, Lebach
  - MorphoSys Research Site, Lübeck
  - MorphoSys Research Site, Mainz
  - MorphoSys Research Site, Münster
  - MorphoSys Research Site, Neustadt
  - MorphoSys Research Site, Oldenburg
  - MorphoSys Research Site, Oldenburg in Holstein
  - MorphoSys Research Site, Potsdam
  - MorphoSys Research Site, Ratingen
  - MorphoSys Research Site, Saarbrücken
  - MorphoSys Research Site, Schorndorf
  - MorphoSys Research Site, Stuttgart
  - MorphoSys Research Site, Villingen-Schwenningen
  - MorphoSys Research Site, Wilhelmshaven
  - MorphoSys Research Site, Wolfsburg
- Italy (23):
  - MorphoSys Research Site, Alessandria
  - MorphoSys Research Site, Ancona
  - MorphoSys Research Site, Aviano
  - MorphoSys Research Site, Bergamo
  - MorphoSys Research Site, Bologna
  - MorphoSys Research Site, Como
  - MorphoSys Research Site, Cremona
  - MorphoSys Research Site, Florence
  - MorphoSys Research Site, Lecce
  - MorphoSys Research Site, Milan
  - MorphoSys Research Site, Modena
  - MorphoSys Research Site, Napoli
  - MorphoSys Research Site, Palermo
  - MorphoSys Research Site, Perugia
  - MorphoSys Research Site, Piacenza
  - MorphoSys Research Site, Ponderano
  - MorphoSys Research Site, Ravenna
  - MorphoSys Research Site, Reggio Calabria
  - MorphoSys Research Site, Rimini
  - MorphoSys Research Site, Roma
  - MorphoSys Research Site, Terni
  - MorphoSys Research Site, Udine
  - MorphoSys Research Site, Vicenza
- South Korea (3):
  - MorphoSys Research Site, Busan
  - MorphoSys Research Site, Seoul
  - MorphoSys Research Site, Ulsan
- Spain (15):
  - MorphoSys Research Site, Badalona
  - MorphoSys Research Site, Barcelona
  - MorphoSys Research Site, L'Hospitalet de Llobregat
  - MorphoSys Research Site, Lugo
  - MorphoSys Research Site, Madrid
  - MorphoSys Research Site, Majadahonda
  - MorphoSys Research Site, Palma de Mallorca
  - MorphoSys Research Site, Pamplona
  - MorphoSys Research Site, Pozuelo de Alarcón
  - MorphoSys Research Site, Sabadell
  - MorphoSys Research Site, Salamanca
  - MorphoSys Research Site, Santander
  - MorphoSys Research Site, Seville
  - MorphoSys Research Site, Valencia
  - MorphoSys Research Site, Valladolid
- Taiwan (3):
  - MorphoSys Research Site, Taichung
  - MorphoSys Research Site, Tainan
  - MorphoSys Research Site, Taipei
- United Kingdom (6):
  - MorphoSys Research Site, Brighton
  - MorphoSys Research Site, Manchester
  - MorphoSys Research Site, Sunderland
  - MorphoSys Research Site, Taunton
  - MorphoSys Research Site, Truro
  - MorphoSys Research Site, Westcliff-on-Sea

REFERENCES:
- [Derived] Nowakowski GS, Yoon DH, Mondello P, Joffe E, Peters A, Fleury I, Greil R, Ku M, Marks R, Kim K, Zinzani PL, Trotman J, Sabatelli L, Waltl EE, Winderlich M, Sporchia A, Kurukulasuriya NC, Cordoba R, Hess G, Salles G. RE-MIND2: comparative effectiveness of tafasitamab plus lenalidomide versus polatuzumab vedotin/bendamustine/rituximab (pola-BR), CAR-T therapies, and lenalidomide/rituximab (R2) based on real-world data in patients with relapsed/refractory diffuse large B-cell lymphoma. Ann Hematol. 2023 Jul;102(7):1773-1787. doi: 10.1007/s00277-023-05196-4. Epub 2023 May 12. PMID 37171597
- [Derived] Nowakowski GS, Yoon DH, Peters A, Mondello P, Joffe E, Fleury I, Greil R, Ku M, Marks R, Kim K, Zinzani PL, Trotman J, Huang D, Waltl EE, Winderlich M, Kurukulasuriya NC, Ambarkhane S, Hess G, Salles G. Improved Efficacy of Tafasitamab plus Lenalidomide versus Systemic Therapies for Relapsed/Refractory DLBCL: RE-MIND2, an Observational Retrospective Matched Cohort Study. Clin Cancer Res. 2022 Sep 15;28(18):4003-4017. doi: 10.1158/1078-0432.CCR-21-3648. PMID 35674661
- See also: Related Info — https://epostersonline.com/soho2021/search/ABCL-346